CLINICAL TRIAL: NCT03199560
Title: A Randomized Controlled Double-blinded Study Comparing the Intraoperative Injection of Lymphatic Mapping Agents Tc 99m Tilmanocept to Tc 99m Filtered Sulfur Colloid in Breast Cancer Patients Undergoing Breast Conservation and Sentinel Lymph Node Biopsy
Brief Title: Tilmanocept vs Sulfur Colloid in Sentinel Lymph Node Biopsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memorial Health University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2016.12.1
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Sentinel Lymph Node Biopsy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Intervention Model Description: double-blinded randomized control trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: A double-blind study. Study compound will be masked before dispensing to care team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tilmanocept (Active Comparator): Tc 99m tilmanocept
  Interventions: Drug: Tc 99m tilmanocept
- Sulfur Colloid (Active Comparator): Tc 99m filtered sulfur colloid
  Interventions: Drug: Tc 99m filtered sulfur colloid

INTERVENTIONS:
Drug: Tc 99m tilmanocept — lymphatic mapping agent
  Other Names: LymphoSeek
  Arms: Tilmanocept
Drug: Tc 99m filtered sulfur colloid — lymphatic mapping agent
  Arms: Sulfur Colloid

SUMMARY:
A randomized controlled double-blinded study comparing the intraoperative injection of lymphatic mapping agents Tc 99m tilmanocept to Tc 99m filtered sulfur colloid in breast cancer patients undergoing breast conservation and sentinel lymph node biopsy

DETAILED DESCRIPTION:
This study is a double-blinded randomized control trial comparing tilmanocept to TSC as intraoperative radiolabeled mapping agents in female patients with early stage breast cancer undergoing partial mastectomy with SLNBx.

To secure this aim, patients who are schedule to undergo partial mastectomy and SLBx will be consented and randomized (randomization table) into one of two experimental arms, tilmanocept or TSC.

These patients will then undergo their scheduled partial mastectomy with SLNBx, with the patient and surgeon blinded to the randomization result.

The respective radiotracers will both be delivered to the OR in the same delivery device and volumes to continue to preserve anonymity of the material. Care will be taken to handle the radiotracers along the standards and guidelines that are already in practice in Memorial Health University Hospital's nuclear medicine department. Two intradermal injections of these radiotracers will be delivered at 3 and 6 o'clock positions at the edge of the areola, after induction of general anesthesia, allowing for less discomfort to the patient.

Methylene blue (5-10 ml) will also be injected in the subareolar space immediately afterwards in all study patients, using a separate syringe, in accordance with the surgeon's current standard practice.

Transcutaneous probing of the axilla measuring counts per second will be performed in 3 minute intervals after injection of the radiotracer. Incision in the axilla can, at the earliest, be at 15 minutes, as this is the FDA approved earliest time for tilmanocept. At this time, if the transcutaneous "hot spot" detected by the gamma detector probe is detected, an incision for SLNBx will proceed. A hot spot is defined as an area of increased radioactivity in the axilla with a fall-off in radioactive counts in adjacent tissue. If a hot spot is not detected, transcutaneous probing will continue at 3 minute intervals until this value is reached. In an effort to not prolong the anesthesia time, incision at 30 minutes will be performed even if a hot spot is not identified transcutaneously.

No changes will be made to the method of SLNBx for this study. As axillary lymph node dissection is no longer the standard of care at the time of SLNBx in partial mastectomy, we will continue the practice of sending the SLN for permanent sectioning, however this will be at the surgeon's discretion. If at the time of surgery there are histologically metastatic nodes or if a sentinel node cannot be identified, the surgeon can proceed to axillary lymph node dissection at their discretion, however for the purposes of this study only SLN data will be tracked (please see below for further information on data collection).

Description of method for SLNBx:

After the intradermal injection of tilmanocept or TSC and sub-areolar injection of methylene blue, and the decision to proceed with SLNBx, the standard incision will be made in the axilla overlying the area with the most counts per second per the gamma probe. The subcutaneous tissues are then dissected to the clavipectoral fascia. The fascia is then incised and the axilla is again probed with the gamma probe. Once a blue node or radioactive node(s) is detected they are excised. A radioactive node will be defined as having counts per second that are 10 times higher than surrounding tissue (background count). Once excised, an "ex-vivo" count will be taken of the sentinel node(s) and recorded. If the background radiation of the axilla is less than 10% the counts per second (cps) of the "hottest" harvested sentinel lymph node, the search for radioactive sentinel nodes will be deemed complete. If there is greater than 10% the counts per second remaining in the axilla, then additional nodes will be identified and excised using the same methods until the background radiation is less than 10% the counts per second of the hottest sentinel nodes removed. Additional nodes which are blue but not radioactive will be excised, as will any clinically suspicious nodes.

ELIGIBILITY:
Inclusion Criteria:

* Women above 18 years of age with biopsy proven, clinically stage 1 or 2 breast cancer who will be undergoing partial mastectomy with SLNBx at Memorial Health

Exclusion Criteria:

* Women under the age of 18,
* Clinically positive axillary nodes
* Neoadjuvant therapy for current breast cancer diagnosis
* Women with previous SLNBx or axillary node dissection
* Pregnant women
* Women with previous radiation above the diaphragm, and below the neck

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-06-22 (Estimated); Study Completion 2019-08-22 (Estimated)

PRIMARY OUTCOMES:
Number of harvested lymph nodes | 1 day
  Looking for differences between the treatment arms in the number of harvest sentinel lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: William Burak, MD, Principal Investigator — Memorial Health University Medical Center
Locations (1):
- Memorial Health University Medical Center, Savannah, Georgia, United States

IPD SHARING:
Plan to Share IPD: No